CLINICAL TRIAL: NCT03957122
Title: Individualized Treatment of Patients With Chronic Tinnitus With Repetitive Transcranial Magnetic Stimulation
Acronym: indiTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of responders in the test sessions was too low.
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Head of Center II and out-patient clinic of the Department of Psychiatry and Psychotherapy, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-820-101
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Tinnitus
Keywords: tinnitus; transcranial magnetic stimulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- individualized rTMS (Experimental): Treatment with the best (highest reduction in tinnitus loudness, most reliable, superior to control condition, most tolerable) protocol as obtained in the test sessions (left vs. right temporoparietal junction, 1Hz, 10Hz, 20Hz, 0.1Hz as active control condition).
  Interventions: Device: repetitive transcranial magnetic stimulation
- standard rTMS in responders (Active Comparator): Treatment with standard protocol: left-sided 1Hz in the group of patients who showed temporary reductions in tinnitus loudness in test sessions.
  Interventions: Device: repetitive transcranial magnetic stimulation
- standard rTMS in non-responders (Active Comparator): Treatment with standard protocol: left-sided 1Hz in the group of patients who did not show temporary reductions in tinnitus loudness in test sessions.
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Stimulation of the temporoparietal junction with repetitive transcranial magnetic stimulation
  * 2000 pulses
  * intensity of 110% resting motor threshold
  * 10 sessions (daily from Monday to Friday)
  * positioning of coil according to EEG position CP5/CP6

SUMMARY:
In the first visit a magnetic resonance imaging measurement will be done for the use of a neuronavigation System with the aim to control for stable coil position over the course of the trial. EEG positions CP5/CP6 will be used for positioning the coil. Two test sessions will examine the temporary reductions in tinnitus loudness after 1Hz, 10Hz, 20Hz and 0.1Hz rTMS as control condition over left and right temporo-parietal junction accompanied by electroencephalography. For the two-week treatment three arms will be evaluated: standard treatment (1Hz left-sided) in the groups with and without temporary reductions in test sessions and the best protocol as elicited in test sessions.

DETAILED DESCRIPTION:
Efficacy of repetitive transcranial magnetic stimulation (rTMS) in chronic tinnitus is moderate. So far single sessions and daily treatment of rTMS were rarely combined. Thus it is not clear if temporary reductions in tinnitus loudness as elicited by short single rTMS sessions can be transferred to daily rTMS treatment. Thus, the aim of the study is to investigate the efficacy and reliability of single sessions of rTMS in chronic tinnitus with respect to temporary reductions in tinnitus loudness accompanied with resting state electroencephalography measurements to investigate the neurophysiological correlates of tinnitus reductions. Two test sessions within one week will be done on the left and right temporoparietal junction using 1Hz, 10Hz, 20Hz and 0.1Hz as active control condition. In the next step patients are divided into three arms with the aim to investigate the efficacy of individualized rTMS. The three arms are 1) patients with temporary tinnitus reductions in test sessions: treatment with the best, most reliable, controlled and most tolerable protocol, 2) patients with temporary tinnitus reductions in test sessions: treatment with 1Hz left-sided rTMS, 3) patients with no temporary tinnitus reductions in test sessions: treatment with 1Hz left-sided rTMS. Treatment will be done for 10 days (Monday - Friday) using 2000 pulses with 110% resting motor threshold. Coil position will be tracked with neuronavigation to ensure stable coil Position over the course of the trial.

ELIGIBILITY:
Inclusion criteria:

* chronic tinnitus (> 6 months)
* at least moderate tinnitus distress
* no or consistent medication
* no or consistent Treatments
* residence in Germany and German speaking

Exclusion Criteria:

* objective tinnitus
* serious and not stable illness (e.g. acute psychosis, severe depression or substance dependence, epilepsy, brain tumor)
* meeting the contraindications for transcranial magnetic stimulation or magnetic resonance imaging (electric devices or metal implants in the body, e.g. cardiac pace maker, insulin pump)
* neurological disorders (e.g. cerebrovascular events, neurodegenerative disorder, epilepsy, brain malformation, severe head trauma)
* addictive disorder with consumption in the last two years
* regular intake of benzodiazepines
* participation in another study parallel to the trial
* pregnancy or breastfeeding period
* psychiatric confinement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
TFI | 2 weeks
  Tinnitus Functional Index

SECONDARY OUTCOMES:
TFI | 12 weeks
  Tinnitus Functional Index
Mini-TQ | 12 weeks
  Tinnitus Questionnaire short version
THI | 12 weeks
  Tinnitus Handicap inventory
Tinnitus Severity | 12 weeks
  Tinnitus numeric Rating scales [0(best) - 10(worst)]
MDI | 12 weeks
  Major Depression Inventory
WHO-QOL BREF | 12 weeks
  Quality of life [4(worst) - 20(best)]
CGI | 12 weeks
  clinical global Impression Change [1(best) - 7(worst)]

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No